CLINICAL TRIAL: NCT02816827
Title: A Randomized, Double Dummy, Double Blind, Placebo Controlled Cross Over Study to Evaluate Efficacy of Investigational Product E-AG-01/ E-AG02/ E-AG-03/ E-AG-04 on Alertness and Mental Fatigue
Brief Title: A Study to Evaluate Efficacy of IP on Alertness and Mental Fatigue
Acronym: ALERMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Enovate Biolife Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: EB/160105/ER/AG
Record Dates: First submitted 2016-03-03; First posted 2016-06-29 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Mental Fatigue
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- E-AG-01 (Experimental): 550 mg of 2 capsules having AG-01 and AG-07 will be administered orally twice daily for one day.
  Interventions: Dietary Supplement: AG-01; Dietary Supplement: AG-07
- E-AG-02 (Experimental): 550 mg of 2 capsules having AG-05 and AG-06 will be administered orally twice daily for one day.
  Interventions: Dietary Supplement: AG-05; Dietary Supplement: AG-06
- E-AG-03 (Experimental): 550 mg of 2 capsules having AG-01 and AG-05 will be administered orally twice daily for one day.
  Interventions: Dietary Supplement: AG-01; Dietary Supplement: AG-05
- E-AG-04 (Experimental): 550 mg of 2 capsules having AG-06 and AG-07 will be administered orally twice daily for one day.
  Interventions: Dietary Supplement: AG-06; Dietary Supplement: AG-07

INTERVENTIONS:
Dietary Supplement: AG-01 — Product to increase mental alertness
  Arms: E-AG-01; E-AG-03
Dietary Supplement: AG-05 — Product to increase mental alertness
  Arms: E-AG-02; E-AG-03
Dietary Supplement: AG-06 — Product to increase mental alertness
  Arms: E-AG-02; E-AG-04
Dietary Supplement: AG-07 — Product to increase mental alertness
  Arms: E-AG-01; E-AG-04

SUMMARY:
The current study is design to asses the effect of E-AG-01/ E-AG-02/ E-AG-03 on mental alertness as compared to placebo.

DETAILED DESCRIPTION:
Intake of caffeinated drinks is known to improve energy levels, alertness, and concentration levels. Caffeine is a stimulant of central nervous system and therefore is probably the most commonly used psychoactive substance in the world. Caffeine intake is preferred by many individuals because moderate amount of caffeine consumption postulates certain beneficial effects on nervous system as well as on general well-being, like increase in the level of alertness and diminution in exhaustion especially in low arousal circumstances (e.g. working at night), improvements in performance on vigilance tasks and simple tasks that require sustained response. Along with these virtues caffeine intake is associated with certain demerits also. High dose of caffeine that is more than 400 mg a day in healthy adults may be associated with adverse events such as psycho motor agitation, insomnia, headache, gastrointestinal complaints depending on several other lifestyle parameters.

Since caffeine intake is habitual, withdrawal of caffeine poses certain concerns on performance like its negative impact on mood levels following its withdrawal.

Hence there is always a need to find an alternative to caffeine which has the same attributes of caffeine but is not associated with its habit forming stance. In order to fulfill this unmet need Enovate Biolife has designed a novel natural caffeine free ingredient which postulates to enhance the mental alertness and combats mental fatigue similar as caffeine without causing adverse effects associated with caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male and female computer literate subjects (able to use computers/related technology efficiently)in the age group of 18-40 years of age.
* Subject should be moderate caffeine consumers.
* All subjects should be predominantly right handed.
* Subject has a body mass index (BMI) of ≥18.5 and <25.00 kg/m2.
* Subjects with Generalized Anxiety Disorder Screener (GAD-7) score ≤ 7.
* Subjects screened for depression by Patient Health Questionnaire-9 (PHQ-9) with score ≤ 14.
* Subjects having score of at least 50 ± 20 two out of three readings on Jin Fan's Attention Network Test (ANT) version 1.3.0 after 24 hrs of caffeine abstinence performed at an interval of 30-60 mins each.
* Subject is willing to refrain from consuming caffeine and caffeine-containing products 24 hrs prior to enrollment and during the study prior to all visit to site.
* Subject agrees to refrain from using turmeric, ginger, cardamom, lemon grass , galangal, beetle leave, and beetle nuts containing products like thai food, tea masala, thai sauces, mouth freshener, paan, etc on the day prior to clinic visit.
* Subject is willing to refrain from vigorous physical activity 12 hrs prior to clinic visit.
* Subject should complete at least 7-8 hours of sleep on the night prior the clinic visit.
* Subject is a non-smoker.
* Female subjects currently in their menstrual period can be included only after the last day of menstrual flow.
* Female Subjects consuming oral contraceptives can be included in study after a washout period of 7 days and are willing to stop its use during the study and opt for barrier contraceptive method.
* Subject understands the study procedures and signed informed consent form to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Subjects unable to abstain from caffeine containing products for 24 hrs.
* Subjects suffering from primary or secondary insomnia with/ without active treatment.
* Subjects with Generalized Anxiety Disorder Screener (GAD-7) score > 7.
* Subjects with Personal health Questionnaire Score > 14.
* Subjects suffering from type II Diabetes Mellitus.
* Subject having health conditions that would prevent him/her from fulfilling the study requirements as judged by the investigator on the basis of medical history and routine laboratory test results.
* Subject has uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the average blood pressure measured at screening as well as randomization.
* Subject has a history or presence of clinically significant cardiac, renal, hepatic, endocrine, pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorders that, in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the subject at undue risk.
* Subject has a history, in the judgment of the investigator, of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Subject has a history or presence of oncological disorders.
* Pregnant/ planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period.
* Use of any psychotropic medication within four weeks of screening and throughout the study.
* Use of antibiotics or signs of active systemic infection. Treatment visits will be rescheduled to allow the subject to wash off of the antibiotic for at least five days prior to any test visit.
* Subject has had exposure to any non-registered drug product within 30 days prior to the screening visit.
* Use of any other dietary supplements or herbal products.
* Recent history of (within 12 months of screening visit 1) or strong potential for alcohol or substance abuse.
* Subject has a known allergy or sensitivity to herbal product(s).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Alertness | Five hours
  To assess the effect on mental alertness by Attention network test after ingestion of single dose of investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Srivastav, M D, Principal Investigator — Enovate Biolife Pvt Ltd
Locations (1):
- Vedic Lifesciences, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brunye TT, Mahoney CR, Lieberman HR, Taylor HA. Caffeine modulates attention network function. Brain Cogn. 2010 Mar;72(2):181-8. doi: 10.1016/j.bandc.2009.07.013. Epub 2009 Sep 5. PMID 19733954
- See also: Caffeine modulates attention network function: BrunyéTT1, Mahoney CR, Lieberman HR, Taylor — http://www.ncbi.nlm.nih.gov/pubmed/19733954